CLINICAL TRIAL: NCT05236478
Title: Efficiency of an Optimized Care Organization for Fatigue Management for Patients With COVID-19.
Acronym: CoviMouv
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN142021/CHUSTE
Record Dates: First submitted 2022-02-10; First posted 2022-02-11 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Fatigue
Keywords: COVID-19; Fatigue; training; therapeutic education; physical activity
MeSH Terms: conditions — COVID-19; Fatigue; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CoviMouv' program: Patients who have benefited from the CoviMouv' program (supervised physical activity program + therapeutic education program) will be included.
  Interventions: Other: CoviMouv' program
- control group: Patients with autonomous physical activity at home or with a community-based physiotherapist will be included. They will have support for the resumption of an adapted physical activity in autonomy, according to the results of the aerobic and anaerobic tests carried out during the initial evaluation (delivery of a training booklet).
  Interventions: Other: Control

INTERVENTIONS:
Other: CoviMouv' program — * An initiation to physical rehabilitation at the hospital center the first week, 3 sessions of 1 hour.
  * A tele-rehabilitation program led by an Adapted Physical Activity (APA) teacher for 3 weeks with 3 sessions of 1 hour per week.
  All the sessions are led by a professional of adapted physical activity and will be personalized and adapted to the functional tests carried out during the initial evaluation.
  * Therapeutic education video-workshops weekly: about (i) the pathophysiology of fatigue in COVID-19, (ii) returning to work, (iii) lifestyle: sleep, physical activity and diet.
  * The medical follow-up will be carried out remotely with 1 weekly teleconsultation with a physiologist.
  * Psychological and / or dietetic follow-up, if necessary, during the program: 1 weekly teleconsultation At the end of the program, each participant is invited to contact the sport-health platform in order to continue the Adapted Physical Activity (APA) practice near home for 2 months.
  Groups: CoviMouv' program
Other: Control — The CoviMouv' program is not presented to theses patients They have support for the resumption of an adapted physical activity in autonomy, according to the results of the aerobic and anaerobic tests carried out during the initial evaluation (delivery of a training booklet).
  Groups: control group

SUMMARY:
Length of hospitalization for COVID-19 infection may be increased due to the persistence of fatigue in 29-46% of cases. Its management is essential to prevent the chronic fatigue . Chronic fatigue syndrome affected between 30 and 40% of patients with SARS in 2003 or MERS in 2005 and persisted beyond 3 years. There is currently no specific treatment for acute or <4 months asthenia. To avoid the transition to chronicity, some authors recommend respecting a long rest period. However, a program combining adapted physical activity and therapeutic patient education has already shown significant benefits for combating recent or semi-recent fatigue following a cardiovascular pathology and even during cancer treatments. Therefore, the existing care pathway for hospitalized patients with COVID-19 was adapted, combining exercise training and therapeutic patient education workshops.

ELIGIBILITY:
Inclusion Criteria:

* Patient living in the Loire region, France
* Patient showing post COVID-19 fatigue (RT PCR positive <1 month)
* Non-intubated patient if hospitalization in intensive care (<72h)
* Patient hospitalized in a Covid unit at the Saint Etienne Hospital

Exclusion Criteria:

* Patient hospitalized in intensive care >72h
* Intubated and ventilated patient in intensive care
* Non-hospitalized patient and community-based medical follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute fatigue post-COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Fatigue evaluation | At 1 Month
  assessed by Chalder Fatigue Scale (CFQ11) with score from 0 to 33. High scores represent high levels of fatigue.

SECONDARY OUTCOMES:
Quality of life (MOS-SF 12) | At 1 Month
  assessed by the medical outcome study short form questionnaire (MOS-SF 12, score from 0 to 100). High scores represent high patient's ability.
Aerobic performances | At 1 Month
  Assessed by the 6-minute walk test (6MWT, walking distance in meter)
Anaerobic performances | At 1 Month
  assessed by the handgrip (muscular strength of biceps in kilogram)
Physical activity | At 1 Month
  assessed by the adult physical activity questionnaire (APAQ, time spend to physical activity in hours/day)
return to work | At 1 Month
  Time needed to return to work (for active workers, time in weeks).
previous activities | At 1 Month
  Time needed to return to previous activities (for retirees, time in weeks).

CONTACTS AND LOCATIONS:
Overall Officials: David HUPIN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No